CLINICAL TRIAL: NCT01971957
Title: Sjogren-Larsson Syndrome: A Longitudinal Study of Natural History, Clinical Variation and Evaluation of Biochemical Markers
Brief Title: Sjogren-Larsson Syndrome: Natural History, Clinical Variation and Evaluation of Biochemical Markers
Acronym: SLS
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0560-12-FB
Record Dates: First submitted 2013-04-30; First posted 2013-10-30 (Estimated); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Sjogren-Larsson Syndrome (SLS)
Keywords: ichthyosis; spasticity; spastic diplegia; intellectual disability
MeSH Terms: conditions — Sjogren-Larsson Syndrome; Ichthyosis; Muscle Spasticity; Cerebral Palsy; Intellectual Disability

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood, urine, skin
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sjogren-Larsson syndrome: There are no cohorts for this study.

SUMMARY:
Sjogren-Larsson syndrome (SLS) is a rare genetic disease in which patients typically exhibit ichthyosis (dry, scaly skin), intellectual disability, spasticity, seizures and a distinctive maculopathy. The purpose of this study is to define the clinical spectrum and natural history of Sjogren-Larsson syndrome, and identify biomarkers that correlate with disease phenotype while establishing a registry for future investigations of biochemical pathogenesis and therapy.

DETAILED DESCRIPTION:
The study will consist of a clinical component and a scientific component consisting of laboratory investigations of potentially useful biochemical (lipid and protein) markers. Up to 50 SLS patients of all ages, gender and ethnic origins will be enrolled. A detailed clinical evaluation will be performed to determine the presence and extent of disease involving the skin, nervous system and eyes. Clinical testing will include brain magnetic resonance imaging (MRI) and spectroscopy (MRS), electroencephalography (EEG), neurocognitive tests, ophthalmologic examination with retinal photographs and optical coherence tomography (OCT), photographs of the skin and tests of cutaneous transepidermal water loss. Laboratory investigations will include lipid analyses (e.g. fatty alcohols, farnesol, fatty acids, ether glycerolipids, etc.) of blood, skin and urine; proteomic analysis of skin (stratum corneum); and measurements of leukocyte fatty alcohol and farnesol oxidation. A skin biopsy (optional) will be obtained for electron microscopy, measurement of lanthanum perfusion (transepidermal water loss), and/or establishing keratinocyte cultures. Correlations between clinical abnormalities and laboratory measurements will be tested to identify the most useful biomarkers for future diagnostic and therapeutic studies. To characterize the progression of phenotypic features over time, patients <6 years of age will be followed yearly and patients ≥6 years of age will be followed every 3 years. In addition, a SLS patient registry will be established as a resource for future investigations in SLS.

ELIGIBILITY:
Inclusion Criteria:

* The only eligibility criterion is that subjects have a genetically or biochemically confirmed diagnosis of Sjogren-Larsson syndrome.

Exclusion Criteria:

* The primary exclusion criteria are the patients' failure to consent or inability to travel to a STAIR site.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will come from cohorts of Sjögren-Larsson syndrome patients currently followed at STAIR sites, from the RDCRN contact registry, and from the pool of new patients who directly contact STAIR sites or are referred to STAIR centers by their physicians.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Characterize the extent and progression of neurocutaneous disease in patients with Sjogren-Larsson syndrome (SLS). | 2017 (up to 5 years)
  Determine the spectrum of clinical disease severity and changes in severity of symptoms over time. Each organ system will be evaluated using validated clinical exams (for example, Modified Ashworth Spasticity Score for neurologic severity) or categorical tests (such as EEG normal or abnormal). The clinical data will be used to develop a quantitative SLS severity score whereby patients will be described (for example, overall severity 1 to 5 with score 1 being the mildest phenotype and score 5 being the most severe). These quantitative outcome measures will be followed over time to assess disease progression.

SECONDARY OUTCOMES:
Identify biomarkers that correlate with disease severity. | 2017 (up to 5 years)
  Blood, urine and skin biomarkers will be explored to identify tests that correlate with clinical severity of SLS. Multiple tests will be performed and outcome measures will be statistically compared to the clinical severity score to determine correlation coefficients, which will be used to establish new biomarkers for SLS.

CONTACTS AND LOCATIONS:
Overall Officials: William B Rizzo, MD, Study Chair — University of Nebraska
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Rizzo WB. Sjogren-Larsson syndrome: molecular genetics and biochemical pathogenesis of fatty aldehyde dehydrogenase deficiency. Mol Genet Metab. 2007 Jan;90(1):1-9. doi: 10.1016/j.ymgme.2006.08.006. Epub 2006 Sep 22. PMID 16996289
- [Background] Lossos A, Khoury M, Rizzo WB, Gomori JM, Banin E, Zlotogorski A, Jaber S, Abramsky O, Argov Z, Rosenmann H. Phenotypic variability among adult siblings with Sjogren-Larsson syndrome. Arch Neurol. 2006 Feb;63(2):278-80. doi: 10.1001/archneur.63.2.278. PMID 16476818
- [Background] Rizzo WB, Craft DA, Somer T, Carney G, Trafrova J, Simon M. Abnormal fatty alcohol metabolism in cultured keratinocytes from patients with Sjogren-Larsson syndrome. J Lipid Res. 2008 Feb;49(2):410-9. doi: 10.1194/jlr.M700469-JLR200. Epub 2007 Oct 30. PMID 17971613
- [Background] Fuijkschot J, Theelen T, Seyger MM, van der Graaf M, de Groot IJ, Wevers RA, Wanders RJ, Waterham HR, Willemsen MA. Sjogren-Larsson syndrome in clinical practice. J Inherit Metab Dis. 2012 Nov;35(6):955-62. doi: 10.1007/s10545-012-9518-6. Epub 2012 Jul 26. PMID 22833178
- [Background] Rizzo WB. The role of fatty aldehyde dehydrogenase in epidermal structure and function. Dermatoendocrinol. 2011 Apr;3(2):91-9. doi: 10.4161/derm.3.2.14619. Epub 2011 Apr 1. PMID 21695018
- [Background] Rizzo WB, Carney G. Sjogren-Larsson syndrome: diversity of mutations and polymorphisms in the fatty aldehyde dehydrogenase gene (ALDH3A2). Hum Mutat. 2005 Jul;26(1):1-10. doi: 10.1002/humu.20181. PMID 15931689
- [Background] Willemsen MA, Van Der Graaf M, Van Der Knaap MS, Heerschap A, Van Domburg PH, Gabreels FJ, Rotteveel JJ. MR imaging and proton MR spectroscopic studies in Sjogren-Larsson syndrome: characterization of the leukoencephalopathy. AJNR Am J Neuroradiol. 2004 Apr;25(4):649-57. PMID 15090362